CLINICAL TRIAL: NCT04331509
Title: COVID-19 Symptom Tracker
Status: Active, not recruiting | Type: Observational
Sponsor: King's College London (Other)
Collaborators: Zoe Global Limited (Other); Massachusetts General Hospital (Other); Harvard School of Public Health (HSPH) (Other); Stanford University (Other)
Responsible Party: Sponsor
Other Study IDs: COVID-19 Symptom tracker
Record Dates: First submitted 2020-03-31; First posted 2020-04-02 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: COVID-19
Keywords: COVID-19; Coronovirus; Symptom tracker; Virus; Pandemic
MeSH Terms: conditions — COVID-19; Virus Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Symptom tracker users: No Intervention
  Interventions: Other: No Intervention

INTERVENTIONS:
Other: No Intervention — No Intervention

SUMMARY:
The viral Covid-19 outbreak is now considered a pandemic according to the World Health Organisation (WHO). A free monitoring app 'COVID-19 Symptom Tracker' has been developed to record and monitor the symptoms of the COVID-19 coronavirus infection; tracking in real time how the disease progresses. The app also records how measures aimed at controlling the pandemic including self-isolation and distancing are affecting the mental health and well-being of participants. The data from the study will reveal important information about the symptoms and progress of COVID-19 infection in different people, and why some go on to develop more severe or fatal disease while others have only mild symptoms do not.

DETAILED DESCRIPTION:
A free monitoring app 'COVID-19 Symptom Tracker' has been developed by health technology company Zoe Global Limited in collaboration with scientists at King's College London, Harvard Medical School, Massachusetts General Hospital and Stanford University. A web-based equivalent is being developed for those unable to download this app. This new app records and monitors the symptoms of COVID-19 coronavirus infection; tracking in real time how the disease progresses. The app also records how measures aimed at controlling the pandemic including self-isolation and distancing affect the mental health and well-being of participants. The app also allows self-reporting where no symptoms are experienced such that it records any users that feel healthy and normal.

The app, has been launched in both the UK and the US. Researchers in other countries are encouraged to obtain the required approvals from Apple and Google to make the app available in their territories.

The data from the study will reveal important information about the symptoms and progress of COVID-19 infection in different people, and why some go on to develop more severe or fatal disease while others have only mild symptoms do not.

It is also hoped that the data generated from this study will help the urgent clinical need to distinguish mild coronavirus symptoms from seasonal coughs and colds, which may be leading people to unnecessarily self-isolate when they aren't infected or inadvertently go out and spread the disease when they are.

Users download the free app COVID-19 Symptom Tracker and record information about their health on a daily basis, including temperature, tiredness and symptoms such as coughing, breathing problems or headaches.

The app is available internationally to the general population and will also be used in two large epidemiological cohorts: The TwinsUK cohort (n=15,000) and Nurses Health Study (n=280,000).

The app will allow scientists to study the spread and development of symptoms across whole populations, both in the UK and abroad, as well as detailed genetic and other studies, particularly with the twins cohort

Any data gathered from the app and study will be used strictly for public health or academic research and will not be used commercially or sold.

ELIGIBILITY:
Inclusion Criteria:

* Adults of 18 years and above, both in the UK and internationally where the app has been approved for download from the Apple App store and Google Play. The web-based equivalent to the app will also be made available via a link for those unable to download.

Exclusion Criteria:

* Anyone below the age of 18; anyone unable to provide informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Anyone who is able to download the app or use the web-based equivalent tool to self-report their symptoms.
Sampling Method: Non-Probability Sample
Enrollment: 10000000 (Estimated)
Dates: Start 2020-03-23 (Actual); Primary Completion 2026-03-23 (Estimated); Study Completion 2026-03-23 (Estimated)

PRIMARY OUTCOMES:
Physical health symptoms | 1 day
  Self reported as physically healthy (tick box)
Lack of physical health symptoms | 1 day
  Self reported as physically not feeling healthy (tick box)

SECONDARY OUTCOMES:
Fever | 1 day
  Self reported remperature (Degrees Celsius)

OTHER OUTCOMES:
Cough | 1 day
  Self reported cough (drop down menu; yes/no)
Fatigue | 1 day
  Self reported fatigue (drop down menu; yes/no)
Headache | 1 day
  Self reported headache (drop down menu; yes/no)
Shortness of breath | 1 day
  Self reported shortness of breath (drop down menu; yes/no)
Sore throat | 1 day
  Self reported sore throat (drop down menu; yes/no)
Loss of smell/ taste | 1 day
  Self reported loss of smell/ taste (drop down menu; yes/no)
Hoarse voice | 1 day
  Self reported hoarse voice (drop down menu; yes/no)
Chest pain or tightness | 1 day
  Self reported chest pain or tightness (drop down menu; yes/no)
Abdominal pain | 1 day
  Self reported abdominal pain (drop down menu; yes/no)
Diarrhoea | 1 day
  Self reported diarrhoea (drop down menu; yes/no)
Confusion | 1 day
  Self reported confusion (drop down menu; yes/no)
Skipping meals | 1 day
  Self reported skipping meals (drop down menu; yes/no)

CONTACTS AND LOCATIONS:
Overall Officials: Tim D Spector, Principal Investigator — King's College London
Locations (2):
- Massachusetts General Hospital, Boston, Massachusetts, United States
- King's College London, London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Access to the COVID-19 Symptom Tracker data will be given to members of the clinical or scientific community as outlined below in accordance with the following privacy policies:
  https://covid.joinzoe.com/privacy-notice
  https://storage.googleapis.com/covid-symptom-tracker-public/privacy-policy-us.pdf
Time Frame: Immediately
Access Criteria: Request to access the COVID-19 Symptom Tracker data should made by submitting an online Data Access Application Form. The form is available on the TwinsUK website.
  https://dtr.eu.qualtrics.com/jfe/form/SV_81U9lmshTofiFeZ
  Decision Process & Outcome:
  Upon submission of the Covid-19 Data Application Form, the TwinsUK data management team will review the application forms received and information on the outcome will be provided within a week. Decisions on the most complex applications will be overseen by the TwinsUK Resource Executive Committee.
  All applicants must belong to the clinical or scientific community, present a valid rationale and must have
  * A healthcare email address
  * An educational email address
  * A track of peer reviewed publications
URL: https://dtr.eu.qualtrics.com/jfe/form/SV_81U9lmshTofiFeZ

REFERENCES:
- [Derived] Lo CH, Nguyen LH, Drew DA, Warner ET, Joshi AD, Graham MS, Anyane-Yeboa A, Shebl FM, Astley CM, Figueiredo JC, Guo CG, Ma W, Mehta RS, Kwon S, Song M, Davies R, Capdevila J, Sudre CH, Wolf J, Cozier YC, Rosenberg L, Wilkens LR, Haiman CA, Marchand LL, Palmer JR, Spector TD, Ourselin S, Steves CJ, Chan AT; COPE Consortium. Race, ethnicity, community-level socioeconomic factors, and risk of COVID-19 in the United States and the United Kingdom. EClinicalMedicine. 2021 Aug;38:101029. doi: 10.1016/j.eclinm.2021.101029. Epub 2021 Jul 17. PMID 34308322
- [Derived] Nguyen LH, Drew DA, Graham MS, Joshi AD, Guo CG, Ma W, Mehta RS, Warner ET, Sikavi DR, Lo CH, Kwon S, Song M, Mucci LA, Stampfer MJ, Willett WC, Eliassen AH, Hart JE, Chavarro JE, Rich-Edwards JW, Davies R, Capdevila J, Lee KA, Lochlainn MN, Varsavsky T, Sudre CH, Cardoso MJ, Wolf J, Spector TD, Ourselin S, Steves CJ, Chan AT; COronavirus Pandemic Epidemiology Consortium. Risk of COVID-19 among front-line health-care workers and the general community: a prospective cohort study. Lancet Public Health. 2020 Sep;5(9):e475-e483. doi: 10.1016/S2468-2667(20)30164-X. Epub 2020 Jul 31. PMID 32745512